CLINICAL TRIAL: NCT04693325
Title: PROlonged Ex-vivo Normothermic Machine PERfusion for Kidney Regeneration
Acronym: PROPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, ipjalwayn, Prof. dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76344
Record Dates: First submitted 2020-06-24; First posted 2021-01-05 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: End Stage Renal Disease
Keywords: normothermic machine perfusion; renal transplantation; kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged normothermic machina perfusion (Experimental): Eligible and consenting patients who will receive a donor kidney will be included for participation in this study. Current practice is to preserve donor kidneys on hypothermic machine perfusion (HMP). In this study, donor kidneys (n=18) will be taken off the HMP after arrival in the transplant center. These will then be perfused with oxygenated perfusate using the NMP device following an optimised NMP protocol.
  Interventions: Procedure: Prolonged normothermic machine perfusion

INTERVENTIONS:
Procedure: Prolonged normothermic machine perfusion — First, a cohort of DCD kidneys (n=6) will be subjected to 1 hour of NMP and subsequently transplanted [NMP1]. Before extending the duration, secondary endpoints will be evaluated. Thereafter, the duration of NMP will be prolonged to 3 hours (n=6) [PNMP3] and consequently 6 hours (n=6) [PNMP6].

SUMMARY:
The investigators would like to introduce and clinically evaluate prolonged normothermic machine perfusion (PNMP) to preserve and assess high-risk donor kidneys prior to transplantation.

DETAILED DESCRIPTION:
Currently kidney transplantation is the only viable option for patients with kidney failure to regain quality of life and health. The number of organs available for transplantation is insufficient with a widening gap between supply and demand. Nowadays, centers accept older and higher risk donor organs with co-morbidity, often leading to non-function, complications and with half of the patients back on dialysis within 15 years. Furthermore, many donor kidneys have to be discarded as too damaged and beyond repair. Increasing the quality and therefore transplantability of these high-risk donor organs could significantly increase the donor kidney pool.

Using prolonged normothermic perfusion of marginal donor organs, the investigators aim to kick start regeneration in the kidney before transplantation, improving function and survival long-term. Furthermore, the choice to accept or decline a donor kidney organ is currently based on subjective criteria and causes great uncertainty amongst clinicians. There is a dire need for tools to aid in decision making and reduce this uncertainty. Biomarkers predictive of graft regeneration are lacking. Samples from perfused kidneys and donor recipients will be collected and analysed to allow the formulation of a kidney fitness index.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing 1st or 2nd kidney transplant
* Patients undergoing a kidney transplantation from DCD Maastricht III & V
* Transplant recipients aged ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Patients undergoing 3rd or subsequent kidney transplant
* Patients undergoing a kidney transplantation from DCD Maastricht I, II & IV
* Transplant recipients aged < 18 years
* Patients receiving multi-organ transplants
* ABO/HLA incompatible transplants
* Highly sensitized patients with a panel-reactive antibody (PRA) ≥85%
* Kidneys with CIT > 12 hrs at the point of arrival at transplant centre
* Kidneys with complex vascular anatomy (≥3 arteries, artery which cannot be can-nulated or attached to the patch holder)
* Kidneys explanted from a donor on normothermic regional perfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
glomerular filtration rate (GFR) | 6 months post transplantation
  renal function defined by the estimated glomerular filtration rate (eGFR) calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

SECONDARY OUTCOMES:
glomerular filtration rate (GFR) | 1 month post transplantation
  renal function defined by the estimated glomerular filtration rate (eGFR) calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
glomerular filtration rate (GFR) | 3 months post transplantation
  renal function defined by the estimated glomerular filtration rate (eGFR) calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
primary non-function | 6 months post transplantation
  defined as permanent lack of graft function from the time of transplantation, was diagnosed when a kidney graft was well perfused (confirmed by ultrasound examination) but never functioned, necessitating dialysis after kidney transplantation
delayed graft function (DGF) | 6 months post transplantation
  defined as the need for postoperative dialysis during the first 7 days after transplantation
patient and graft survival | 6 months post transplantation
  time from transplant to patient death, and graft failure
adverse events | 6 months post transplantation
  defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the normothermic machine perfusion of the donor kidney prior to transplantation
postoperative complications | 6 months post transplantation
  graded according to the comprehensive complication index

CONTACTS AND LOCATIONS:
Overall Officials: Ian PJ Alwayn, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: No